CLINICAL TRIAL: NCT01508884
Title: Efficacy and Effectiveness of Intradermal Trivalent Influenza Vaccine With Topical Imiquimod, a Double Blind Randomized Controlled Trial
Brief Title: Intradermal Trivalent Influenza Vaccine With Imiquimod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HKU-2012-432
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Illness
Keywords: intradermal; influenza; vaccination
MeSH Terms: conditions — Chronic Disease; Influenza, Human | interventions — Influenza Vaccines; Imiquimod; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IM vaccine and placebo cream (Active Comparator): A single dose of intramuscular influenza vaccine (15ug non-adjuvanted 2011/2012 TIV) with pre-treatment of the injected skin with aqueous cream
  Interventions: Biological: influenza vaccine; Drug: Aqueous cream
- ID vaccine and placebo cream (Active Comparator): A single dose of intradermal influenza vaccine (15ug non-adjuvanted 2011/2012 TIV) with pre-treatment of the injected skin with aqueous cream
  Interventions: Biological: influenza vaccine; Drug: Aqueous cream
- ID vaccine and imiquimod cream (Experimental): A single dose intradermal influenza vaccine (15ug non-adjuvanted 2011/2012 TIV) with pre-treatment of the injected skin with imiquimod cream applied to the skin before vaccination
  Interventions: Biological: influenza vaccine; Drug: Imiquimod

INTERVENTIONS:
Biological: influenza vaccine — single dose of intradermal 15 mcg non-adjuvanted 2011/2012 trivalent influenza vaccine
  Other Names: Intanza 15
  Arms: ID vaccine and imiquimod cream
Drug: Imiquimod — pretreatment with topical imiquimod cream to the injection site before vaccination
  Other Names: Aldara
  Arms: ID vaccine and imiquimod cream
Biological: influenza vaccine — single dose of intradermal 15mcg non-adjuvanted 2011/2012 trivalent influenza vaccine
  Other Names: Intanza 15
  Arms: ID vaccine and placebo cream
Drug: Aqueous cream — pretreatment with topical aqueous cream to the injection site before vaccination
  Arms: ID vaccine and placebo cream
Biological: influenza vaccine — single dose of intramuscular 15mcg non-adjuvanted 2011/2012 trivalent influenza vaccine
  Other Names: Vaxigrip
  Arms: IM vaccine and placebo cream
Drug: Aqueous cream — pretreatment with topical aqueous cream to the injection site before vaccination
  Arms: IM vaccine and placebo cream

SUMMARY:
Despite the WHO International Health Regulations Emergency Committee declared an end to the 2009 H1N1 pandemic globally, the emergence of the novel 2009 H1N1 virus in March 2009 has affected more than 214 countries with at least 18000 deaths [1]. Patients with chronic underlying illness and extreme of ages are at risk of developing severe disease and complications [2-3]. Resistance to oseltamivir has also been reported [4]. Therefore, vaccination with the 2010/2011 trivalent influenza vaccine (TIV) with the 2009 H1N1-like virus incorporated will be the best protection against the influenza infection, especially among the at risk population. Recent study on dose sparing seasonal influenza vaccine delivered via a novel intradermal microneedle has demonstrated good immunogenic responses similar to full-dose intramuscular vaccination [6]. Poor immunogenicity of the H1N1 2009 component of the trivalent influenza has been reported [7].

Study has also suggested the combined intradermal vaccination with local stimulation of dermal antigen presenting cells by applying imiquimod cream (Aldara) to the injection site, which activate antigen presenting cells (APC) through the toll-like receptor 7 (TLR7) may produce better immunogenicity [8].

Imiquimod cream is currently registered for the treatment of warts and basal cell carcinoma. Scientific evidence has demonstrated that after treatment with imiquimod, the antigen is processed and presented to cells of the adaptive immune system leading to clearance of the virus and subsequent clearance of the lesions [9]. In addition to functional maturation, imiquimod induces migration of dendritic cells from the dermis to draining lymph nodes [10,11]. Subcutaneous administration of imiquimod as vaccine adjuvant simultaneously with the antigen of interest, has shown to induce enhanced responses towards the administered antigen [12].

We therefore performed a prospective, double blind, randomized controlled study to compare the safety and immunogenicity between intradermal 2011/2012 TIV immunization with pretreatment of imiquimod cream and conventional full dose intramuscular 2011/2012 TIV immunization with pretreatment of aqueous cream as control.

DETAILED DESCRIPTION:
References

1. World Health Organization. Influenza A (H1N1) - update 95 [cited 2010 April 10]. Available from http://www.who.int/csr/don/2009_12_30/en/index.html
2. Echevarria-Zuno S, Mejia-Arangure JM, Mar-Obeso AJ, et al. Infection and death from influenza A H1N1 virus in Mexico: a retrospective analysis. Lancet 2009; 374: 2072-9.
3. Louie JK, Acosta M, Winter K, et al. Factors associated with death or hospitalization due to pandemic 2009 influenza A(H1N1) infection in California. JAMA 2009; 302: 1896-902.
4. Jain S, Kamimoto L, Bramley AM, et al. Hospitalized patients with 2009 H1N1 influenza in the United States, April-June 2009. N Engl J Med 2009; 361:1935-44.
5. Chen H, Cheung CL, Tai H, et al. Oseltamivir-resistant influenza A pandemic (H1N1) 2009 virus, Hong Kong, China. Emerg Infect Dis 2009;15:1970-2.
6. Van Damme P, Oosterhuis-Kafeja F, Van der Wielen M, et al. Safety and efficacy of a novel microneedle device for dose sparing intradermal influenza vaccination in healthy adults. Vaccine 2009;27:454-9
7. Myers CA, Faix DJ, Blair PJ. Possible reduced effectiveness of the 2009 H1N1 component of live, attenuated influenza vaccine. Clin Infect Dis. 2011;15;53:207-8.9.
8. Roukens R, Vossen AC, Boland GJ, et al. Intradermal hepatitis B vaccination in non-responders after topical application of imiquimod (Aldara). Vaccine 2010;4288-4293.
9. Tyring S, Conant M, Marini M, Van Der Meijden W, Washenik K. Imiquimod, an international update on therapeutic uses in dermatology. Int J Dermatol 2002;41(11):810-6.
10. Burns Jr RP, Ferbel B, Tomai M, Miller R, Gaspari AA. The imidazoquinolines, imiquimod and R-848, induce functional, but not phenotypic, maturation of human epidermal Langerhans' cells. Clin Immunol 2000;94(1):13-23.
11. Suzuki H, Wang B, Shivji GM, Toto P, Amerio P, Tomai MA, et al. Imiquimod, a topical immune response modifier, induces migration of Langerhans cells. J Invest Dermatol 2000;114(1):135-41.
12. Thomsen LL, Topley P, Daly MG, Brett SJ, Tite JP. Imiquimod and resiquimod in a mouse model: adjuvants for DNA vaccination by particle-mediated immunotherapeutic delivery. Vaccine 2004;22(13-14):1799-809.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients at the age of 21 or above with chronic illness and given written informed consent
* Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

* Clinically significant immune-related diseases or significant recent co-morbidities
* Inability to comprehend and to follow all required study procedures
* History or any illness that might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Have received 2011/2012 TIV
* Have a recent history (documented, confirmed or suspected) of a flu-like disease within a week of vaccination.
* Have a known allergy to eggs or other components of the Study Vaccines (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein), or history of any anaphylaxis, serious vaccine reactions, to any excipients.
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination, or women who are breastfeeding.
* Female of childbearing potential, not using any acceptable contraceptive methods for at least 2 months prior to study entry or that do not plan to use acceptable birth control measures during the first 3 weeks after vaccination.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long-term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed).
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Have known active human immunodeficiency virus (HIV) infection, acute hepatitis B or C infection, autoimmune hepatitis and related cirrhosis
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.
* History of progressive or severe neurological disorders
* Have received any licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination (only exception being unadjuvanted seasonal influenza vaccines which are allowed until 1 week prior to and after 1 week study vaccinations).
* Axillary temperature ≥ 38°C or oral temperature ≥ 38.5°C within 3 days of intended study vaccination
* Surgery planned during the study period that in the Investigator's opinion would interfere with the study visits schedule
* Have a history of alcohol or drug abuse in the last 5 years.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | day 7
  The percentage of subjects with an hemagglutination inhibition antibody titre <10 at baseline and a post-vaccination titre of ≥40 or a titre >10 at baseline and at least a four-fold increase in titre post-vaccination on day 7

SECONDARY OUTCOMES:
Geometric mean titer old increase in influenza antibody titer | day 21
  The GMT fold increase in influenza antibody titer by hemagglutination inhibition or microneutralization antibody assays on day 21 compared to day 0
Seroprotection rate | day 21
  The percentage of subjects achieving an antibody titer achieving an influenza antibody titer of 1:40 or above by hemagglutination inhibition or microneutralization antibody assay on day 21
Adverse events (Immediate) | 30 minutes after vaccination
  Patients who develop systemic or local adverse events within 30 minutes of vaccination
Geometric mean titer old increase in influenza antibody titer | day 7
  The GMT fold increase in influenza antibody titer by hemagglutination inhibition or microneutralization antibody assay on day 7 compared to day 0
Seroprotection rate | day 7
  The percentage of subjects achieving an antibody titer achieving an influenza antibody titer of 1:40 or above by hemagglutination inhibition or microneutralization antibody assay on day 7
Geometric mean titer old increase in influenza antibody titer | year 1
  The GMT fold increase in influenza antibody titer by hemagglutination inhibition or microneutralization antibody assay at year 1 compared to day 0
Seroprotection rate | year 1
  The percentage of subjects achieving an antibody titer achieving an influenza antibody titer of 1:40 or above by hemagglutination inhibition or microneutralization antibody assay at year 1
Seroconversion rate | Year 1
  The percentage of subjects with an hemagglutination inhibition antibody titre <10 at baseline and a post-vaccination titre of ≥40 or a titre >10 at baseline and at least a four-fold increase in titre post-vaccination at year 1
Adverse events (7 days) | 7 days after vaccination
  Patients who develop systemic or local adverse events within 1 week of vaccination
Seroconversion rate | Day 21
  The percentage of subjects with an hemagglutination inhibition antibody titre <10 at baseline and a post-vaccination titre of ≥40 or a titre >10 at baseline and at least a four-fold increase in titre post-vaccination on day 21
Geometric mean titer old increase in influenza antibody titer | Day 14
  The GMT fold increase in influenza antibody titer by hemagglutination inhibition or microneutralization antibody assay at year 1 compared to day 0
Seroprotection rate | Day 14
  The percentage of subjects achieving an antibody titer achieving an influenza antibody titer of 1:40 or above by hemagglutination inhibition or microneutralization antibody assay at year 1
Seroconversion rate | Day 14
  The percentage of subjects with an hemagglutination inhibition antibody titre <10 at baseline and a post-vaccination titre of ≥40 or a titre >10 at baseline and at least a four-fold increase in titre post-vaccination at year 1
Effectiveness | 1 year post vaccination
  hospitalization for pneumonia or influenza
Effectiveness | 1 year post vaccination
  Nasopharyngeal sample positive for influenza A

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong